CLINICAL TRIAL: NCT05454449
Title: Effect of Dynamic Taping on Landing Biomechanical Characteristics in Volleyball and Basketball Players With Symptoms of Patellar Tendinopathy - Motor Control and Biomechanical Characteristics During the Landing Task
Brief Title: Effect of Dynamic Taping on Landing Biomechanics in Athletes With Symptoms of Patellar Tendinopathy
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, National Yang Ming Chiao Tung University
Other Study IDs: YM109067F(2)
Record Dates: First submitted 2022-07-02; First posted 2022-07-12 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Biomechanical Phenomena
Keywords: patellar tendinopathy; volleyball; basketball; landing; biomechanics; EMG; muscle activation; kinetics; kinematics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- symptomatic group: Individuals with patellar tendon pain last for 3 months Individuals age between 18-40 years old Individuals had trained in volleyball or basketball for more than two years Individuals still played volleyball or basketball for at least 90 minutes a week Victorian Institute of Sport Assessment (VISA) Questionnaire score ≦80
- asymptomatic group: Individuals without any lower extremity pain(NRS>3/10) in past 3 months Individuals age between 18-40 years old Individuals had trained in volleyball or basketball for more than two years Individuals still played volleyball or basketball for at least 90 minutes a week Victorian Institute of Sport Assessment (VISA) Questionnaire score >80

SUMMARY:
Patellar tendinopathy (PT) is an overuse injury associated with loading activities, and popular among basketball and volleyball players. Although altered biomechanical characteristics during landing has been suggested as one of the risk factors for the development of PT, previous evidence failed to show the link between the sagittal plane biomechanics of the hip and knee joint and PT; and little was known about the frontal and horizontal plane biomechanics in athletes with PT. While other factors such as motor control or muscle activation also have not been explored fully. The purpose of this study is to compare hip motor control and biomechanical characteristics of the hip and knee joint during landing in athletes with and without symptomatic PT.

DETAILED DESCRIPTION:
Background: Patellar tendinopathy is an overuse injury associated with loading activities, and it is thought to be caused by repetitive force applied to the patellar tendon. Patellar tendinopathy is popular among basketball and volleyball players, particularly in men. Although altered biomechanical characteristics during landing has been suggested as one of the risk factors for the development of patellar tendinopathy, previous evidence failed to show the link between the sagittal plane biomechanics of the hip and knee joint and patellar tendinopathy; and little was known about the frontal and horizontal plane biomechanics in athletes with patellar tendinopathy. Among those factors contributing to the biomechanical characteristics, hip and quadriceps strength were shown linked with the presence of patellar tendinopathy, while other factors such as motor control or muscle activation have not been explored fully. The purpose of this study is to compare hip motor control and biomechanical characteristics of the hip and knee joint during landing in athletes with and without symptomatic patellar tendinopathy. The investigators hypothesize that the athletes with symptomatic patellar tendinopathy have poorer motor control and different landing biomechanics as compared with asymptomatic athletes.

Method: the investigators plan to recruit seventeen symptomatic patellar tendinopathy athletes for the experimental group, using demographic data (sex, age, height, weight, exercise type) of experimental group to match seventeen non-symptomatic athletes as control group. The assessment included hip motor control in various directions, and measurement of kinetics, kinematics and muscle activation during the step-down task, drop vertical jump and countermovement jump using the computer-aided video motion analysis system (Vicon) and the surface EMG (Noraxon). The group difference will be tested using t-test for the motor control ability and biomechanical characteristics. The significant level was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* at the age of 18 to 40 years old
* volleyball and basketball players have more than 2 years training experience
* over 90 minutes of training time per week

symptomatic group:

* having patellar tendon pain during loading task last for 3 months
* VISA-P questionnaire score ≦80

asymptomatic group:

* without any lower extremity pain(NRS3/10) in past 3 months
* VISA-P questionnaire score >80

Exclusion Criteria:

* Underwent sports physical therapy for knee pain in the past three months.
* Currently have any other chronic or acute lower limb injuries with a pain score >3/10.
* Self-reported pregnancy.
* Had surgery, fractures, or received steroid injections for the patellar tendon in the lower limbs.
* with a history of rheumatoid arthritis, systematic and neurological diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * 18 to 40 years old volleyball and basketball players
  * Volleyball and basketball players with more than 2 years' training experience
  * Volleyball and basketball players train over 90 minutes per week
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Fen Shih, Ph.D, Study Director — Department of Physical Therapy and Assistive Technology, National Yang-Ming Chiao-Tung University
Locations (1):
- National Yang-Ming Chiao-Tung University, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Taipei and New Taipei City via social media between February 2023 and June 2023. The first participant was enrolled on February 13, 2023 and the last participant was enrolled in June 2023
Period: Overall Study
Arm/Group | Symptomatic Group | Asymptomatic Group
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symptomatic Group | Asymptomatic Group | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 17 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 174.07 (7.71) | 174.03 (8.40) | 174.05 (7.822)
Specializing in [Count of Participants; unit: Participants]
  volley ball | 13 | 13 | 26
  basketball | 4 | 4 | 8
Dominal leg [Count of Participants; unit: Participants]
  right | 16 | 16 | 32
  left | 1 | 1 | 2
Body weight [Mean (Standard Deviation); unit: kg] | 68.59 (8.89) | 68.69 (8.56) | 68.64 (8.46)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.73 (2.29) | 22.64 (1.55) | 22.68 (1.89)
Training time per week [Mean (Standard Deviation); unit: min/wk] | 442.94 (228.85) | 425.29 (301.91) | 434.71 (259.48)
VISA-PCh [Mean (Standard Deviation); unit: units on a scale] — The VISA-PCh scale is a validated Chinese version questionnaire designed to assess the severity of patellar tendinopathy, commonly known as jumper's knee.
  Questionnaire consists of eight questions, covering three key areas: Pain, Function and Sports Participation.
  Each question is scored, with a total possible score from 0-100. A higher score indicates better tendon health and lower symptom severity, while a lower score suggests more significant impairment due to patellar tendinopathy.
  units on a scale | 64.12 (10.16) | 93.06 (5.98) | 78.59 (16.68)
Jumping height [Mean (Standard Deviation); unit: cm] | 63.84 (10.79) | 64.46 (9.94) | 64.15 (10.38)
Height of spike jump [Mean (Standard Deviation); unit: cm] | 72.29 (12.19) | 72.21 (11.66) | 72.25 (11.93)
Ankle DF ROM in weight bearing [Mean (Standard Deviation); unit: degrees]
  Right side | 36.61 (6.82) | 37.24 (4.80) | 36.92 (5.73)
  Left side | 39.90 (4.64) | 38.90 (4.28) | 39.40 (4.36)
Hip extensor power [Mean (Standard Deviation); unit: percentage of body weight]
  Right side | 44.93 (10.73) | 43.39 (11.08) | 44.16 (10.61)
  Left side | 46.71 (11.64) | 43.53 (9.64) | 45.12 (10.49)

OUTCOME MEASURES:

1. Primary Outcome: Hip Flexion Angles
Description: Measure the hip joint angle when the knee reaches the maximum flexion angle during the landing phase of the countermovement jump
Time Frame: In the experiment, the maximum knee flexion during the landing phase of the countermovement jump
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Symptomatic Group | Asymptomatic Group
Number analyzed (Participants) | 17 | 17
degrees | 86.59 (15.51) | 73.65 (20.05)
Statistical Analysis 1: Comparison: Symptomatic Group vs Asymptomatic Group; Test type: Other; p = 0.047, t-test, 2 sided

2. Primary Outcome: Maximal Knee Flexion Angle
Description: In the countermovement jump test, the force received by the force plate changes from 0 to a positive value during the landing phase. Measure the maximal knee flexion angle during this phase.
Time Frame: The landing phase of the countermovement jump in the experiment
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Symptomatic Group | Asymptomatic Group
Number analyzed (Participants) | 17 | 17
degrees | 97.87 (15.17) | 83.70 (14.21)
Statistical Analysis 1: Comparison: Symptomatic Group vs Asymptomatic Group; Test type: Other; p = 0.009, t-test, 2 sided

3. Primary Outcome: Hip Abduction Angle
Description: Measure the hip abduction angle when the knee reaches the maximum flexion angle during the landing phase of the countermovement jump
Time Frame: In the experiment, the maximum knee flexion during the landing phase of the countermovement jump
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Symptomatic Group | Asymptomatic Group
Number analyzed (Participants) | 17 | 17
degrees | 13.97 (6.50) | 10.68 (3.76)
Statistical Analysis 1: Comparison: Symptomatic Group vs Asymptomatic Group; Test type: Other; p = 0.082, t-test, 2 sided

4. Primary Outcome: Knee Joint Flexion Angle
Description: Perform the step-down test on a 15 cm high table to measure the knee flexion angle of the foot on the table when the side foot is at the lowest point.
Time Frame: the contralateral foot is at its lowest point in step-down test in the experiment
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Symptomatic Group | Asymptomatic Group
Number analyzed (Participants) | 17 | 17
degrees | 60.79 (5.57) | 65.18 (5.05)
Statistical Analysis 1: Comparison: Symptomatic Group vs Asymptomatic Group; Test type: Other; p = 0.022, t-test, 2 sided

5. Primary Outcome: Motor Control Ability
Description: Having 4 motor control tests:
  Hip Flexion Control: Maintain an upright posture in a single-leg small knee bend. The knee aligns with the 2nd toe in the sagittal plane and >5 cm beyond the toes.
  Internal/External Rotation Control:Perform a single-leg small knee bend while rotating the pelvis and upper body toward the opposite/same side. Rotate 35°/30° without excessive L/E compensation.
  Hip Adduction Control:Maintain a single-leg stance with symmetrical shoulders and pelvis. Pelvic lateral displacement <10 cm, left-right displacement difference <2 cm.
  Scoring Criteria:
  Avoid uncontrolled movements, perform isolated movements correctly, achieve adequate ROM, maintain normal breathing, control movements in eccentric/concentric phases, execute smoothly, stay relaxed and aware, ensure fluid transitions, avoid compensations, complete without feedback/support, and show no fatigue.
  Total score range: 0-52, converted to a percentage for comparison(0-100%).
Time Frame: during the experiment, up to 4 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptomatic Group | Asymptomatic Group
Number analyzed (Participants) | 17 | 17
score on a scale | 78 (11) | 86 (8)
Statistical Analysis 1: Comparison: Symptomatic Group vs Asymptomatic Group; Test type: Other; p = 0.016, t-test, 2 sided

6. Secondary Outcome: Maximum Muscle Activity of Biceps Femoris
Description: Before the task, the subjects were asked to prone on the bed with their hips at 0 degrees and tested knee at 45 degrees of flexion, and to do isometric contractions with the utmost strength. The muscle contraction signals were recorded by EMG, and the average value of five measurements was taken as maximal voluntary contraction (MVC) of biceps femoris.
  The countermovement jump test requires the participant to cross their arms over the chest, squat down, and then jump as high as possible before landing. The landing phase is identified when the ground reaction force recorded by the force plate transitions from zero to a positive value. Using a trigger, the force plate data is synchronized with EMG data to determine the peak activation of the biceps femoris muscle during the landing phase.
  The biceps femoris contraction signals collected during the task were divided by the maximum biceps femoris contraction signal, and the results were standardized for comparison between individuals.
Time Frame: Immediately during the experiment
Measure: Mean (Standard Deviation); unit: percentage of MVC
Arm/Group | Symptomatic Group | Asymptomatic Group
Number analyzed (Participants) | 17 | 17
percentage of MVC | 16.03 (7.50) | 21.44 (6.02)
Statistical Analysis 1: Comparison: Symptomatic Group vs Asymptomatic Group; Test type: Other; p = 0.029, t-test, 2 sided

7. Secondary Outcome: Muscle Activity of Biceps Femoris
Description: Before the task, the subjects were asked to prone on the bed with their hips at 0 degrees and tested knee at 45 degrees of flexion, and to do isometric contractions with the utmost strength. The muscle contraction signals were recorded by EMG, and the average value of five measurements was taken as maximal voluntary contraction (MVC) of biceps femoris.
  The countermovement jump test requires the participant to cross their arms over the chest, squat down, and then jump as high as possible before landing. The landing phase is identified when the GRF recorded by the force plate transitions from zero to a positive value. Using a trigger, the force plate data and kinematics data is synchronized with EMG data to determine the activation of the biceps femoris muscle during maximal knee flexion in the landing phase.
  The signals collected during the task were divided by the maximum biceps femoris contraction signal, and the results were standardized for comparison between individuals.
Time Frame: Immediately during the experiment
Measure: Mean (Standard Deviation); unit: percentage of MVC
Arm/Group | Symptomatic Group | Asymptomatic Group
Number analyzed (Participants) | 17 | 17
percentage of MVC | 4.93 (1.89) | 7.40 (2.91)
Statistical Analysis 1: Comparison: Symptomatic Group vs Asymptomatic Group; Test type: Other; p = 0.007, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: during the experiment, up to 4 hours
Description: no any adverse event
Arm/Group | Symptomatic Group | Asymptomatic Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT05454449/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT05454449/ICF_001.pdf